CLINICAL TRIAL: NCT03958838
Title: Peer Support to Enhance the Shanghai Integration Model of Diabetes Care: Dissemination to 12 Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Merck Foundation (Unknown)
Responsible Party: Principal Investigator, Weiping Jia, Professor, Director of Shanghai Diabetes Institute, Shanghai 6th People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-028
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Type2 Diabetes; PreDiabetes
Keywords: Peer Support; Social Support; Primary Care; Integrated Care; Community-Based; Self-Management; Diabetes Care
MeSH Terms: conditions — Prediabetic State | interventions — Primary Health Care

STUDY DESIGN:
Intervention Model Description: Intervention group and Control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Subjects will receive usual care from community health center staff. In addition, they will also receive a variety of community-level and individual-level interventions, categorized broadly into three levels.
  At the community level, subjects will receive the 5 Key Diabetes Messages that Everyone Should Know and the 6 Modules of Basic Diabetes Education. At the individual level, subjects and their families will be invited to participate in group activities, co-organized by community health staff, CHC staff, and CSMG peer leaders. Subjects will receive in-person peer support through these group activities, with follow up through telephone calls and text messaging. For subjects that have poorly controlled diabetes or are experiencing emotional distress related to their diabetes, CSMG peer leaders will work closely with them to help them solve problems around their diabetes.
  Interventions: Behavioral: Peer Support Integrated with Primary Care
- Control Group (No Intervention): Subjects in the control group will receive usual care from community health center staff.

INTERVENTIONS:
Behavioral: Peer Support Integrated with Primary Care — Peer leaders will deliver support that address the four key functions of peer support, providing 1) assistance in daily self-management, 2) linkages to clinical care and community resources, 3) social and emotional support, and 4) ongoing, flexible support over time.
  Arms: Intervention Group

SUMMARY:
This project will disseminate a community-level intervention that integrates peer support from Community Self-Management Groups (CSMGs) and primary care through Community Health Centers (CHC). The model and program materials were developed and refined from the first year of implementation within community health centers in Shanghai. This project will be implemented in 12 communities in 6 districts across Shanghai, representing a diverse cross section of the population. A total of 1440 subjects will be recruited from the 12 intervention communities and 720 control subjects will be recruited from 4 control communities.

DETAILED DESCRIPTION:
The development of contemporary diabetes care offers new hope for long and satisfying lives of those with the disease, but also provides increased challenges for integration across the many dimensions of care (varied medications in addition to insulin, specialty services, diet, physical activity, stress management, etc.) and across the many who contribute to care (specialists, primary care providers, nurses, dietitians and patient educators, family members, friends, worksites). The Shanghai Integration Model (SIM) has made great strides to integrating specialty/hospital care with primary/community care. The addition of peer support can enhance patient engagement within that integrated care. Peer support can also integrate care with the daily behaviors and patterns that optimal diabetes management requires and with the family members and others in individuals' daily lives who can support diabetes management.

This project will disseminate a community-level intervention that integrates peer support from Community Self-Management Groups (CSMGs) and primary care through Community Health Centers (CHC). The model and program materials were developed and refined from the first year of implementation within community health centers in Shanghai. This project will be implemented in 12 communities in 6 districts across Shanghai, representing a diverse cross section of the population. A total of 1440 subjects will be recruited from the 12 intervention communities and 720 control subjects will be recruited from 4 control communities.

The program is a collaboration among the Shanghai Sixth People's Hospital, Shanghai Jiao Tong University, the Shanghai Diabetes Institute, the National Office for Primary Diabetes Care, the Shanghai Municipal Health Commission, the Shanghai Municipal Center for Disease Control and Prevention, and, at the University of North Carolina-Chapel Hill, Peers for Progress, widely recognized for its leadership in promoting peer support in health care and prevention.

Collaborators:

Shanghai Sixth People's Hospital Shanghai Jiao Tong University Shanghai Diabetes Institute National Office for Primary Diabetes Care Shanghai Municipal Health Commission Shanghai Municipal Center for Disease Control and Prevention University of North Carolina at Chapel Hill, Peers for Progress

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥ 18
* Chinese
* Has type 2 diabetes or prediabetes
* Patient at participating CHC

  • Intervention group: 120 subjects at each of 12 CHCs
* ~40 patients (Pre-diabetes including IFG or IGT)
* ~40 patients (Diabetics with poor control, FPG≥9.7 mmol/L)
* ~40 patients (Newly-diagnosed diabetics within 2 years)

  • Control group: 240 control subjects at each of 2 CHCs (Yichuan and Zhaoxiang) and 120 control subjects at each of 2 CHCs (Xuhang and Waigang)

  o (Yichuan and Zhaoxiang)
* ~80 patients (Pre-diabetes including IFG or IGT)
* ~80 patients (Diabetics with poor control, FPG≥9.7 mmol/L)
* ~80 patients (Newly-diagnosed diabetics within 2 years)

  o (Xuhang and Waigang)
* ~40 patients (Pre-diabetes including IFG or IGT)
* ~40 patients (Diabetics with poor control, FPG≥9.7 mmol/L)
* ~40 patients Newly-diagnosed diabetics within 2 years)

Exclusion Criteria:

- No serious mental illness (i.e. major depression, schizophrenia, bipolar disorder, obsessive compulsive disorder, panic disorder, post-traumatic stress disorder, borderline personality disorder)

Withdrawal criteria:

- No longer a patient at participating CHC (moved, deceased, extended hospitalization)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2160 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline HbA1c and at 12 months | Baseline, 12 months
  HbA1c (%)

SECONDARY OUTCOMES:
Change from Baseline Fasting Blood Glucose and at 12 months | Baseline, 12 months
  FPG (mmol/L)
Change from Baseline Blood Pressure and at 12 months | Baseline, 12 months
  SBP and DBP (mmHg)
Change from Baseline BMI and at 12 months | Baseline, 12 months
  Height (cm) and weight (kg)
Change from Baseline Blood Lipids and at 12 months | Baseline, 12 months
  Total cholesterol, triglycerides, HDL, LDL (mmol/L)
Change from Baseline Waist circumference and at 12 months | Baseline, 12 months
  Waist circumference (cm)
Change from Baseline Hemoglobin and at 12 months | Baseline, 12 months
  Hemoglobin (g/L)
Change from Baseline Red Blood Cell Count and at 12 months | Baseline, 12 months
  Red blood cell count (10^12/L)
Change from Baseline Mean Corpuscular Volume and at 12 months | Baseline, 12 months
  Mean Corpuscular Volume (fL)
Change from Baseline Mean Corpuscular Hemoglobin and at 12 months | Baseline, 12 months
  Mean Corpuscular Hemoglobin (pg)
Change from Baseline Liver Functioning and at 12 months | Baseline, 12 months
  ALT (U/L), AST (U/L), Alkaline phosphatase (U/L), r-GT (U/L)
Change from Baseline Bilirubin and at 12 months | Baseline, 12 months
  Total bilirubin (μmol/L), Direct bilirubin (μmol/L)
Change from Baseline Blood Urea and at 12 months | Baseline, 12 months
  Blood urea (mmol/L)
Change from Baseline Serum Creatinine and at 12 months | Baseline, 12 months
  Serum creatinine (μmol/L)
Change from Baseline Uric Acid and at 12 months | Baseline, 12 months
  Uric acid (μmol/L)
Change from Baseline Urine Albumin/Creatinine Ratio and at 12 months | Baseline, 12 months
  Albumin (mg/L), Creatinine (mmol/L)
Change in Insulin Functioning at 6 and 12 months | Baseline, 12 months
  Insulin (pmol/L)
Change in C-peptides at 6 and 12 months | Baseline, 12 months
  C-peptide (nmol/L)
Change in CRP at 6 and 12 months | Baseline, 12 months
  CRP (mg/dL）
Change from Baseline Diabetes Self Care Behaviors and 12 months | Baseline, 12 months
  9 items from Summary of Diabetes Self Care Activities and Behavioral Risk Factor Surveillance System. Items 1-7 measure diabetes self care activities during the previous 7 days. Items 1, 2, 4-7 are assessed on a scale of 0 to 7 days. Item 3 is assessed on scale of 1-4, where 1 represents very low levels of daily activity and 4 represents very high levels of daily activity. Items 8 and 9 are yes/no questions that measure cigarette intake over the past 7 and 30 days.
Change from Baseline General Quality of Life and 12 months | Baseline, 12 months
  6-item EQ-5D, a standardized instrument for measuring generic health status. The respondents are asked to choose one of the statements which best describes their health status on the surveyed day. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions). Item 6 is the visual analogue scale, in which respondents are asked to mark their health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100, where 0 corresponds to "the worst health you can imagine", and 100 corresponds to "the best health you can imagine"
Change from Baseline Diabetes Quality of Life and 12 months | Baseline, 12 months
  4-item Diabetes Distress Scale, an abbreviated version of the 17-item Diabetes Distress Scale. The respondents are asked to respond to which degree each of the items has bothered them in the past month on a 6-point scale (1-6), where 1 is not a brother and 6 is very bothersome. Scores are summed and divided by 4 to calculate the mean. Mean scores of 3 or higher (moderate distress) are considered worthy of clinical attention.
Change from Baseline Depression and 12 months | Baseline, 12 months
  8-item Patient Health Questionnaire (PHQ), the PHQ-9 minus the last question on suicidal thoughts. The PHQ is a standard instrument used in primary care settings to screen for the presence and severity of depression. The respondents are asked how often they have been bothered by each of the 8 items in the past 2 weeks on a 4 point scale (0-3), where 0 is "not all" and 3 is "nearly every day". The scores for each item are summed to produce a total score between 0 and 24 points. A total score of 0 to 4 represents no significant depressive symptoms. A total score of 5 to 9 represents mild depressive symptoms; 10 to 14, moderate; 15 to 19, moderately severe; and 20 to 24, severe.
Change from Baseline Insulin Attitudes and 12 months | Baseline, 12 months
  ITAS items, 6 questions
Change in Neighborhood Interactions and 12 months | Baseline, 12 months
  6 questions
Change in Peer Support Engagement and Health Care Utilization and 12 months | Baseline, 12 months
  5 questions

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Jia, MD, PhD, Principal Investigator — Shanghai 6th People's Hospital; Edwin B Fisher, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (16):
- China (16):
  - Anting Huangdu Community Health Center, Shanghai, Shanghai Municipality
  - Baihe Community Health Center, Shanghai, Shanghai Municipality
  - Dachang Qilian Community Health Center, Shanghai, Shanghai Municipality
  - Fangsong Community Health Center, Shanghai, Shanghai Municipality
  - Guangzhong Community Health Center, Shanghai, Shanghai Municipality
  - Huamu Community Health Center, Shanghai, Shanghai Municipality
  - Liantang Community Health Center, Shanghai, Shanghai Municipality
  - Luodian Community Health Center, Shanghai, Shanghai Municipality
  - Nanxiang Community Health Center, Shanghai, Shanghai Municipality
  - Nicheng Community Health Center, Shanghai, Shanghai Municipality
  - Ouyang Community Health Center, Shanghai, Shanghai Municipality
  - Waigang Community Health Center, Shanghai, Shanghai Municipality
  - Xiao Kunshan Community Health Center, Shanghai, Shanghai Municipality
  - Xuhang Community Health Center, Shanghai, Shanghai Municipality
  - Yichuan Community Health Center, Shanghai, Shanghai Municipality
  - Zhaoxiang Community Health Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher EB, Boothroyd RI, Coufal MM, Baumann LC, Mbanya JC, Rotheram-Borus MJ, Sanguanprasit B, Tanasugarn C. Peer support for self-management of diabetes improved outcomes in international settings. Health Aff (Millwood). 2012 Jan;31(1):130-9. doi: 10.1377/hlthaff.2011.0914. PMID 22232103
- [Background] Zhong X, Wang Z, Fisher EB, Tanasugarn C. Peer Support for Diabetes Management in Primary Care and Community Settings in Anhui Province, China. Ann Fam Med. 2015 Aug;13 Suppl 1(Suppl 1):S50-8. doi: 10.1370/afm.1799. PMID 26304972
- [Background] Chan JC, Sui Y, Oldenburg B, Zhang Y, Chung HH, Goggins W, Au S, Brown N, Ozaki R, Wong RY, Ko GT, Fisher E; JADE and PEARL Project Team. Effects of telephone-based peer support in patients with type 2 diabetes mellitus receiving integrated care: a randomized clinical trial. JAMA Intern Med. 2014 Jun;174(6):972-81. doi: 10.1001/jamainternmed.2014.655. PMID 24781960
- [Derived] Evans M, Liu Y, Wu X, Cai C, Tang PY, Maggy Coufal M, Qian Y, Fisher EB, Jia W. Community organization guides standardization, adaptability, and innovation: lessons from peer support in the Shanghai Integration Model. Transl Behav Med. 2023 Aug 11;13(8):519-532. doi: 10.1093/tbm/ibac094. PMID 37406180